CLINICAL TRIAL: NCT06666010
Title: A Registered Clinical Trial of PEX010-Assisted Therapy for Stimulant Use Disorder: A Safety, Feasibility and Efficacy Study
Brief Title: PEX010-Assisted Therapy for Stimulant Use Disorder: A Safety, Feasibility and Efficacy Study
Acronym: PATSUD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Filament Health Corp. (Industry)
Collaborators: University of British Columbia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PATSUD_F
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Stimulant Use Disorder

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Adult participants with confirmed StUD - Active (Experimental): PEX010 containing 25 mg psilocybin
  Interventions: Drug: PEX010-Assisted Therapy
- Adult participants with confirmed StUD - Placebo (Placebo Comparator): PEX010 containing 1 mg psilocybin
  Interventions: Drug: PEX010(01)

INTERVENTIONS:
Drug: PEX010-Assisted Therapy — The investigational medicinal product PEX010, containing 25 mg psilocybin, is a capsule for oral administration that contains the drug substance PYEX.
  Arms: Adult participants with confirmed StUD - Active
Drug: PEX010(01) — The investigational medicinal product PEX010(01), containing 1 mg psilocybin, is a capsule for oral administration that contains the drug substance PYEX.
  Arms: Adult participants with confirmed StUD - Placebo

SUMMARY:
The goal of this clinical trial is to learn if PEX010 is effective for the treatment of Stimulant Use Disorder in adults. The study will also assess the safety and feasibility of administering PEX010 to this population. The main questions it aims to answer are:

Does PEX010 reduce stimulant use?

What medical problems do participants experience when taking PEX010?

Researchers will compare an active PEX010 dose containing 25 mg psilocybin to an active placebo arm, to see if PEX010 works to reduce stimulant use.

Participants will:

Take PEX010 or the active placebo once during the study, engage in cognitive behavioural therapy, and visit the clinic twice weekly for study intervention and follow-up assessments.

DETAILED DESCRIPTION:
In this randomized, controlled trial study participants will receive one capsule of PEX010 containing 25 mg or 1 mg of psilocybin, in conjunction with therapy.

Following screening and baseline visits, participants will receive 2 preparation sessions, 1 PEX010 dosing session, 1 integration session, and 7 follow-up visits.

ELIGIBILITY:
Inclusion Criteria:

* Are between 19 and 65 years old.
* Have signed the informed consent form for the study
* Have moderate to severe amphetamine stimulant use disorder (ASUD) as determined by the Mini-International Neuropsychiatric Interview (MINI 7.0.1), and clinical review by the study physician. The focus will be on illicit methamphetamine use.
* Are treatment-seeking but not currently receiving other treatments for SUD.
* Have stable housing.
* Have a local support person (close friend or family member) that is available to accompany them home from the study drug session.
* Are of non-childbearing potential and/or using adequate contraception methods as defined by Health Canada.
* Non-childbearing potential is defined as (i) self-reported postmenopausal status (12 months of spontaneous amenorrhea and ≥ 45 years of age); or (ii) documented surgical sterilization
* Have a negative pregnancy test at screening and prior to the study drug session. Must agree to use adequate contraception through 10 days after the study drug session. Adequate contraception methods include intrauterine devices, oral hormones plus barrier contraception, abstinence, injectable or implanted hormonal methods, or vasectomized/non-sperm carrying sole partner. Barrier methods alone are not considered effective methods of contraception.
* Be willing to refrain from caffeine for ≥12 hours, cannabis and stimulants for ≥24 hours, and all other drugs for ≥5 days prior to PEX010 administration such that there are no clinical signs of intoxication or withdrawal.
* Able and willing to follow study procedure.
* Able to understand and communicate in English.
* Complete the Columbia Suicide Severity Rating Scale (CSSRS)
* Results from safety laboratory tests (CBC, AST and ALT, TSH, HbA1c) are within normal limits.

Exclusion Criteria:

* Are experiencing or at risk for significant withdrawal.
* Have any medical condition that would be contraindicated, including previously diagnosed conditions:
* seizure disorder or history of seizures;
* a history of significantly impaired hepatic function;
* a history of unstable or uncontrolled cardiovascular disease (coronary artery disease, heart failure, clinically significant ECG abnormality);
* uncontrolled hypertension, resting blood pressure > 140/90 mmHg; baseline prolongation of QTc interval: >450 ms in both males and females;
* a history of major central nervous system disease (history of cerebrovascular accident, masses, aneurysm);
* a history of uncontrolled obstructive airway disease or significant respiratory compromise;
* a history of uncontrolled thyroid disease;
* a history of uncontrolled insulin dependent diabetes that may preclude safe participation in the study;
* a history of narrow-angle glaucoma;
* gastrointestinal conditions which may affect psilocybin absorption (i.e. stenosing peptic ulcer, pyloroduodenal obstruction);
* a history of active obstructive urological conditions (i.e. symptomatic prostatic hypertrophy, bladder-neck obstruction) that may preclude safe participation in the study.
* Have a personality disorder deemed to be high risk (antisocial, borderline, narcissistic) assessed via the SCID-5-PD.
* Have a personal history or family history of either mania/hypomania or psychosis, including substance-induced psychosis.
* Have any history of Hallucinogen Perception Disorder
* Have a history of suicide attempt within the last 6 years or a suicidal ideation in the last year.
* Are currently taking medications with known interactions with psilocybin (e.g., antidepressants, antipsychotics)
* Are pregnant, breastfeeding, or not using adequate contraceptives if of childbearing potential.
* Any other finding(s) based on the screening process that the investigator determines makes the candidate unsuitable for the study
* Results from safety laboratory tests (CBC, AST and ALT, TSH, HbA1c) are not within normal limits
* Have baseline heart rate outside of normal limits (e.g., >100 beats per minute).
* Subjects currently on medications with serotonergic activity, or taking inhibitors of UGT1A9, UGT1A10, MAO and aldehyde or alcohol dehydrogenase.

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Estimated)
Dates: Start 2025-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Changes in Amphetamine-type Stimulant Use | 3 Months
  The difference between treatment and active placebo groups in the proportion of subjects abstinent from illicit methamphetamine use over the course of the 3-month assessment period assessed by Timeline Followback (TLFB) and urine drug tests (UDT).

SECONDARY OUTCOMES:
Number of AEs and SAEs | 3 Months
  Total number of adverse events (AEs) and serious adverse events (SAEs) reported during the 3-month assessment period.

IPD SHARING:
Plan to Share IPD: Undecided